CLINICAL TRIAL: NCT05468281
Title: RAFF5 Proposal: Project to Improve the Quality and Safety of the Immediate and Subsequent Care of Patients Seen in the Emergency Department With Acute Atrial Fibrillation and Flutter
Brief Title: RAFF5 Proposal: Improve the Quality and Safety of Patients Seen in the Emergency Department for Acute Atrial Fibrillation and Flutter
Acronym: RAFF5
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 3875
Record Dates: First submitted 2022-05-25; First posted 2022-07-21 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: Safety; Emergency Department; Management guidelines
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before Period: The before period (12 months) serves as the control period prior to implementation; data will be collected by health records review.
- After Period: The after period (12 months) will be when patients are prospectively enrolled, and outcomes assessed.
  Interventions: Other: Checklist implementation

INTERVENTIONS:
Other: Checklist implementation — . Our strategies will include a) selection of local physician champions from the ED and cardiology; b) discussion of the goals of the study with the local physician groups; c) formal introduction of the CAEP Checklist to the physicians and nurses by means of presentations at staff meetings, emails, and an online video; d) development of an action plan to address local barriers to implementation; e) creation of a free smartphone application; f) regular reminders; and g) and distribution of charts of site compliance.
  Groups: After Period

SUMMARY:
Acute atrial fibrillation (AF) and flutter (AFL) are the most common arrhythmias requiring management in the emergency department (ED). They are characterized by sudden onset of a rapid heart rate which may be irregular (AF) or regular (AFL). Our focus is on episodes of acute AF or AFL which are usually less than 48 hours in duration and are highly symptomatic, requiring rapid treatment in the ED. Management guidelines for acute AF/AFL have changed substantially in recent years with several recent revisions published by the Canadian Cardiovascular Society (CCS) and the Canadian Association of Emergency Physicians (CAEP). The 2021 CAEP Acute Atrial Fibrillation/Flutter Best Practices Checklist (CAEP Checklist) was very recently published to assist ED physicians in Canada and elsewhere manage patients who present to the ED with acute AF/AFL (Figure 1).

The overall goal of this project is to improve the quality and safety of the immediate and subsequent care of patients seen in the ED with acute AF and AFL by implementing the principles of the CAEP Checklist at both The Ottawa Hospital (TOH) EDs and by working with TOH cardiologists to provide rapid cardiology follow-up processes for patients discharged from the ED. The Investigators propose a before-after cohort study using an interrupted time series design to evaluate implementation involving 720 patients at the two TOH EDs over a 24-month period.

ELIGIBILITY:
Inclusion Criteria:

* include all eligible patient visits to the participating EDs during the study period regardless of how they are managed.
* include stable patients aged 18 and over,
* presenting with an episode of acute AF or AFL of at least 3 hours duration,
* where symptoms require ED management by rhythm or rate control.

Exclusion Criteria:

* The study will exclude patients who have any of:

  1. permanent AF;
  2. deemed unstable and required immediate electrical cardioversion; or
  3. primary presentation was for another condition rather than arrhythmia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting to the emergency department with Atrial Fibrillation (AF) or Atrial Flutter (AFL).
Sampling Method: Probability Sample
Enrollment: 1108 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Improve the quality and safety of ED management of AF and AFL | 14 day
  the quality and safety of ED management based upon the CAEP Checklist management. best practices. The study team will use a score sheet which will identify specific managements for AF and AFL that are 1) optimal; 2) suboptimal; 3) unsafe.

SECONDARY OUTCOMES:
Use of cardioversion (chemical or electrical) in the ED | Duration of the ED visit, approximately 4-12 hours.
use of rate control and the final heart rate at disposition | Duration of the ED visit, approximately 4-12 hours.
prescription of OAC on discharge | Duration of the ED visit, approximately 4-12 hours.
  Whether or not they were given an outpatient prescription for oral anticoagulants in accordance with the 2021 CAEP Checklist
consultations done in the ED by cardiology | Duration of the ED visit, approximately 4-12 hours.
  Whether or not the patient had an (unnecessary) consultation done in the ED by cardiology
Adverse events attributable to medical management | Duration of the ED visit, approximately 4-12 hours.
  adverse events including: i) conduction problems; ii) dysrhythmias; iii) hypotension requiring treatment; iv) respiratory events; f) admission to a hospital unit; and g) use of the rapid referral process.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Stiell, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Plan to share data at the end of the study will be reviewed on a case by case basis.

REFERENCES:
- [Derived] Stiell IG, Taljaard M, Beanlands R, Johnson C, Golian M, Green M, Kwok E, Brown E, Nemnom MJ, Eagles D. RAFF-5 Study to Improve the Quality and Safety of Care for Patients Seen in the Emergency Department With Acute Atrial Fibrillation and Flutter. Can J Cardiol. 2024 Sep;40(9):1554-1562. doi: 10.1016/j.cjca.2024.01.037. Epub 2024 Feb 7. PMID 38331027